CLINICAL TRIAL: NCT00534846
Title: The Effect of Toremifene Treatment to the Magnetic Resonance Imaging Findings in Women Suffering From Premenstrual Mastalgia
Brief Title: The Effect of Toremifene Treatment to the Magnetic Resonance Imaging (MRI) Findings in Premenstrual Mastalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Satakunta Central Hospital (Other)
Collaborators: Tampere University (Other)
Responsible Party: Sinikka Oksa, Satakunta Central Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: tore20mg; EudraCT 2006-006109-97
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2009-05-13 (Estimated); Status verified 2009-05

CONDITIONS: Breast Pain
Keywords: premenstrual syndrome; mastalgia; toremifene; selective estrogen receptor modulators
MeSH Terms: conditions — Mastodynia; Premenstrual Syndrome | interventions — Toremifene; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A placebo (Placebo Comparator): The participants were randomly allocated to receive toremifene (20 mg) or placebo during the luteal phase for three consecutive menstrual cycles.
  Interventions: Drug: placebo
- B toremifene (Active Comparator): The participants were randomly allocated to receive toremifene (20 mg) or placebo during the luteal phase for three consecutive menstrual cycles.
  Interventions: Drug: toremifene

INTERVENTIONS:
Drug: toremifene — The medication is given in tablet form, and the participants are instructed to take one tablet daily from cycle day 15 until the next menstruation. The active (toremifene 20 mg) and control (placebo) tablets were identical in appearance.
  Other Names: magnetic resonance imaging; cyclic breast pain
  Arms: B toremifene
Drug: placebo — tablet equal to toremifene, one tablet daily from cycle day 15 to menstruation during three cycles
  Arms: A placebo

SUMMARY:
The purpose of this study is to determine the effect of toremifene treatment to the MRI findings of the breast in women suffering from premenstrual mastalgia.

DETAILED DESCRIPTION:
Benign breast pain is a common complaint of women in western countries. As many as 41-69% of women reported having mastalgia sufficient to interfere with their daily routines. Approximately 8-10% of premenopausal women suffer monthly from moderate to severe breast pain.Tamoxifen has previously been found to be effective in reducing premenstrual mastalgia. We showed that another triphenylethylene derivative, toremifene, significantly alleviated cyclical breast pain as compared to placebo. In this study women suffering from cyclical breast pain are randomly allocated to receive toremifene (20mg) or placebo during the luteal phase for three consecutive cycles. The patients are then crossed over after a wash-out period to placebo or toremifene, respectively. The MRI investigations are made at two occasions during the premenstrual period after three cycles of toremifene and after three cycles of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Premenstrual mastalgia
* Age 20-45 years
* Reliable non-hormonal contraception

Exclusion Criteria:

* Pregnancy
* Breast cancer or uterine corpus cancer
* Unexplained menstrual disorders
* Serious health problems
* Hormonal contraception, including hormonal IUD trade name Mirena
* Oestrogen and/or progestin treatment
* Hysterectomy and/or oophorectomy or radiation therapy
* Artificial cardiac pacemaker/metallic prostheses

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
the effects to the MRI findings | after three cycles toremifene and placebo plus wash-out cycle, seven months
magnetic resonance imaging changes | seven months

SECONDARY OUTCOMES:
cyclic breast pain relief, quality of life, acceptability of treatment | seven months
breast pain | seven months

CONTACTS AND LOCATIONS:
Overall Officials: SINIKKA OKSA, MD, Principal Investigator — Satakunta Central Hospital; JOHANNA MÄENPÄÄ, Study Director — Tampere University Hospital
Locations (1):
- Satakunta Central hospital, department of gynaecology and obstetrics, Pori, Finland

REFERENCES:
- [Background] Oksa S, Luukkaala T, Maenpaa J. Toremifene for premenstrual mastalgia: a randomised, placebo-controlled crossover study. BJOG. 2006 Jun;113(6):713-8. doi: 10.1111/j.1471-0528.2006.00943.x. PMID 16709215